CLINICAL TRIAL: NCT06273748
Title: Retrospective and Prospective Observational Study on Non-infectious Chronic Uveitis in Pediatric Age
Brief Title: RChildUV:Study on Non-infectious Chronic Uveitis in Pediatric Age
Status: Recruiting | Type: Observational
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Gabriele Simonini, Head of Rheumatology, Meyer Children's Hospital IRCCS
Other Study IDs: RChildUV
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Uveitis is an inflammatory disease of the uvea, one of the highly vascularized fundamental structures of the eye. It is a rare condition in children, with an incidence in the pediatric population ranging from 2% to 14% of all uveitis cases. The diagnosis and management of patients with uveitis rely on a multidisciplinary approach involving an ophthalmologist, a rheumatologist, and an infectious disease specialist to establish the correct diagnosis and assess the involvement of other organs. In Italy, there is no national or regional registry for non-infectious chronic uveitis as per the Prime Ministerial Decree (DPCM) of March 3, 2017 (Identification of surveillance systems and registries for mortality, tumors, and other diseases). However, many clinical centers adopt data recording systems to evaluate the quality of care and to study diseases and outcomes. The Universitary Hospital Meyer Institute Research Hospital (IRCCS) is a national referral center for managing these pediatric cases of non-infectious chronic uveitis, estimated to constitute 95% of all pediatric uveitis cases

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-infectious chronic uveitis before the age of 16;
* signed informed consent form.

Exclusion Criteria:

* Patients with a diagnosis of infectious uveitis
* history of malignant pathology,
* history of demyelinating pathology,
* history of cerebral vasculitis

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The data of patients who have been under the care of the hospital since 2010 will be included, and new patients diagnosed from the date of Ethical Committee approval onwards for the next 10 years will also be included
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2032-02-01 (Estimated); Study Completion 2032-05-02 (Estimated)

PRIMARY OUTCOMES:
Describe a population of paediatric patients with chronic non-infectious uveitis | thorugh the study and after 1 year
  * Frequency of each aetiology of uveitis
  * Frequency of signs and symptoms at onset of uveitis
  * Frequency of laboratory findings
  * Frequency of each anatomical subtype of uveitis
Describe a population of paediatric patients with chronic non-infectious uveitis | 6 months, 12 months, 2 years and then every year
  * Frequency of complications at onset, 6 months, 12 months, 2 years, then every year
  * Frequency of impaired visual acuity (LogMAR0.4-1) and blindness (LogMAR>=1) at onset and at different time points (6 months, 12 months, 18 months, 2 years, then every year)
Identify any differences between the different forms of uveitis in terms of characteristics and outcomes | thorugh the study and after 1 year
  * Frequency of complications and impaired visual acuity
  * Description of laboratory characteristics
Identify risk factors for a more severe course | thorugh the study and after 1 year
  Percentages of children with impaired visual acuity
  * Percentages of children with ocular complications
Frequency achievement of response for each drug according to the definition of response | thorugh the study and after 1 year
  Frequency achievement of response for each drug according to the definition of response of the MIWGUC group
Time to archieve the response after drug initiation | thorugh the study and after 1 year
  Time to archieve the response after drug initiation
Achievement of inactive disease on therapy according to the definition of MIWGUC | thorugh the study and after 1 year
  Achievement of inactive disease on therapy according to the definition of MIWGUC
Time to achieve inactive disease on therapy according to the definition of MIWGUC | thorugh the study and after 1 year
  Time to achieve inactive disease on therapy according to the definition of MIWGUC
Presence and percentages of flares on therapy after achievement of remission on therapy | thorugh the study and after 1 year
  Presence and percentages of flares on therapy after achievement of remission on therapy
Time to the first flare on therapy | thorugh the study and after 1 year
  Time to the first flare on therapy
Time to flare after drug withdrawal | 6, 12 and 18 months, 2 years then every year
  Time to flare after drug withdrawal
  * Proportion of Flare after drug withdrawal in general at the last available follow-up
  * Proportion of children who flared after drug withdrawal at 6, 12 and 18 months, 2 years then every year

CONTACTS AND LOCATIONS:
Locations (5):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States
- - ATTIKON General Hospital, Athens, Greece
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence, Firenze
  - Ospedale Spedali Civili di Brescia, Brescia
  - IRCCS materno infantile Burlo Garofolo, Trieste

IPD SHARING:
Plan to Share IPD: No